## NCT07211698

## A QUALITATIVE STUDY EXPLORING ETHNIC MINORITIES' EXPERIENCES OF HEALTHCARE INTERVENTIONS DELIVERED AT HOME OR IN COMMUNITY CENTRES

Ethnic Minorities' Experiences of Healthcare Intervention

27 OCTOBER 2025





## **INFORMED CONSENT FORM (VERBAL)**

| Version 3.0, 27.10.2025 | |
|-------------------------|---------------------|
| REC ref: FMHS 212-0725 | Participant number: |

Chief Investigator: Dr Katie Robinson

After describing the study to the participant, the researcher must discuss the following statements, and the participant will provide verbal consent (i.e. say yes) to take part in the study.

Please write 'yes' on the box to confirm.

| 1. | Do you confirm that you understood the information sheet version 3.0 dated 27.10.2025, provided and explained to you for the qualitative study and have had the opportunity to ask questions? |
|---|---|
| 2. | Do you understand that your participation is voluntary and that you are free to withdraw at any time? |
| 3. | Do you understand that the results of the interview may be looked at by someone not part of the study team to check that the study is being carried out correctly as required by UK law? |
| 4. | Do you understand that even if you withdraw from the above study, any data collected about you up until this point will be kept and used in the final analysis? |
| 5. | Do you consent to the use of an interpreter, direct quotes, fieldnotes, audio recording and transcription of the interview? |
| 6. | Do you consent to the storage of your personal information for the purposes of this study including on a computer? |
| 7. | Do you understand that any information that could identify you will be kept confidential and no personal information will be included in the study report or other publications? |
| 8. | Do you agree not to disclose anything that has been discussed during the study conversations outside of the study? |
| 9. | Do you agree to take part in the study? |



| Optional | |
|---|---|
| 10. | Do you consent for the researcher to have contact information about you to get in touch with what the study found? |
| | Do you consent for the researcher to contact you to take part in future research study? |
| | 2. Are you happy for the researcher to use your postcode for deprivation index that means checking whether where people live have any influence on the healthcare intervention delivered to them at home or in community centres? |

| to them at home or in community centres? | | |
|------------------------------------------|------------------------|------|
| Participants contact details | | |
| Name: | | |
| Telephone: | | |
| Email: | | |
| Postcode <b>NOT</b> your full address: | | |
| Name of researcher | Researcher's signature | Date |



## FOR WITNESS OR INTERPRETER/TRANSLATOR USE ONLY

Complete this section if participant is not able to read the study information and/or sign for themselves but has capacity to give consent OR if the study information has been interpreted or translated to the participant.

| WITNESS STATEMENT: | | |
|---|---|---|
| I witnessed accurate reading of the consent form to the potential participant, who could ask any questions and received satisfactory answers | | |
| I confirm that participant gave their consent freely. | | |
| Witness | Signature | Date |
| First Name and Surname<br>(BLOCK CAPITALS) | 0.9 | |
| INTERPRETER/TRANSLATOR STATEMENT: | | |
| I was present during the meeting between the researcher Joy Watterson and the participant. I translated/ interpreted information for the participant. | | |
| I confirm that study information was interpreted/ translated accurately. | | |
| Interpreter/translator | Signature | Date |
| First Name and Surname<br>(BLOCK CAPITALS) | | |